CLINICAL TRIAL: NCT00001076
Title: A Phase I Safety and Immunogenicity Trial of Live Recombinant Canarypox ALVAC-HIV (vCP205) and HIV-1 SF-2 rgp120 in HIV-1 Uninfected Volunteers to Evaluate Accelerated Vaccine Schedules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 029; 10579 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity; Avipoxvirus; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: ALVAC-HIV MN120TMG (vCP205)
Biological: ALVAC-RG Rabies Glycoprotein (vCP65)
Biological: rgp120/HIV-1 SF-2

SUMMARY:
To evaluate the safety and immunogenicity of an accelerated schedule of recombinant canarypox vaccine ALVAC-HIV MN120TMG (vCP205) versus control followed by boost with rgp120/HIV-1 SF2 vaccine in HIV-negative volunteers.

Frequent injections of ALVAC-HIV vCP205 may result in more rapid induction of cytotoxic T-lymphocytes. This trial will evaluate whether an accelerated vaccination schedule can produce immunological responses comparable to those obtained in other trials of ALVAC-HIV vCP205.

DETAILED DESCRIPTION:
Frequent injections of ALVAC-HIV vCP205 may result in more rapid induction of cytotoxic T-lymphocytes. This trial will evaluate whether an accelerated vaccination schedule can produce immunological responses comparable to those obtained in other trials of ALVAC-HIV vCP205.

Volunteers are randomized to receive immunization with either ALVAC-HIV vCP205 or ALVAC-RG rabies glycoprotein (vCP65) at days 0, 7, 14, and 21, followed by boost with rgp120/HIV-1 SF2 at days 28 and 84. A third cohort receives ALVAC-HIV vCP65 on the same schedule followed by boost with placebo.

ELIGIBILITY:
Inclusion Criteria

Volunteers must have:

* Normal history and physical exam.
* Negative ELISA and Western blot for HIV.
* CD4 count >= 400 cells/mm3.
* Normal urine dipstick with esterase and nitrite.
* Lower-risk sexual behavior.

Exclusion Criteria

Co-existing Condition:

Volunteers with the following symptoms or conditions are excluded:

* Positive hepatitis B surface antigen.
* Medical or psychiatric condition (such as recent suicidal ideation or present psychosis) that precludes compliance.
* Occupational responsibilities that preclude compliance.
* Active syphilis. NOTE: Subjects with serology documented to be a false positive or due to a remote (> 6 months) treated infection are eligible.
* Active tuberculosis. NOTE: Subjects with a positive PPD and a normal chest x-ray showing no evidence of TB and not requiring isoniazid therapy are eligible.
* Allergy to egg products or neomycin.
* Occupational exposure to birds.

Volunteers with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, autoimmune disease, or use of immunosuppressive medications.
* History of anaphylaxis or other serious adverse reactions to vaccines.
* Prior immunization against rabies.
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension).
* Prior psychiatric condition (such as history of suicide attempts or past psychosis) that precludes compliance.
* History of cancer unless there has been surgical excision that is considered to have achieved cure.

Prior Medication:

Excluded:

* Live attenuated vaccines within 60 days prior to study entry. NOTE: Medically indicated killed or subunit vaccines (e.g., influenza, pneumococcal) do not exclude if administered at least 2 weeks from HIV immunizations.
* Experimental agents within 30 days prior to study entry.
* Prior HIV vaccines.
* Prior rabies immunization.

Prior Treatment:

Excluded:

* Blood products or immunoglobulin within 6 months prior to study entry. Identifiable high-risk behavior for HIV infection, such as
* injection drug use within past 12 months.
* higher- or intermediate-risk sexual behavior.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34
Dates: Study Completion 1997-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belshe R, Study Chair
Locations (3):
- United States (3):
  - UAB AVEG, Birmingham, Alabama
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Univ. of Rochester AVEG, Rochester, New York

REFERENCES:
- [Background] Corey L, Weinhold K, Montefiori D, McElrath J, Excler JL, Duliege AM, Stablein D. Combination candidate HIV vaccines using a canarypox vector (vCP205) followed by boosting with gp120(SF-2). Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:209 (abstract no LB18)
- [Background] Evans T, Corey L, Clements-Mann ML, Weinhold K, Belshe RB, Excler JL, Duliege AM. CD8+ CTL induced in AIDS vaccine evaluation group phase I trials using canarypox vectors (ALVAC) encoding multiple HIV gene products (vCP125, vCP205, vCP300) given with or without subunit boost. Int Conf AIDS. 1998;12:277 (abstract no 495/21192)
- [Background] Bender TJ, Tang J, Rivers C, Mulligan MJ, Kaslow RA. Grouping by HLA class I supertype does not enhance HLA associations with CTL responses to ALVAC-HIV canarypox vaccine components. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 193)
- [Background] Belshe RB, Gorse GJ, Mulligan MJ, Evans TG, Keefer MC, Excler JL, Duliege AM, Tartaglia J, Cox WI, McNamara J, Hwang KL, Bradney A, Montefiori D, Weinhold KJ. Induction of immune responses to HIV-1 by canarypox virus (ALVAC) HIV-1 and gp120 SF-2 recombinant vaccines in uninfected volunteers. NIAID AIDS Vaccine Evaluation Group. AIDS. 1998 Dec 24;12(18):2407-15. doi: 10.1097/00002030-199818000-00009. PMID 9875578
- [Background] Sabbaj S, Mulligan MJ, Hsieh RH, Belshe RB, McGhee JR. Cytokine profiles in seronegative volunteers immunized with a recombinant canarypox and gp120 prime-boost HIV-1 vaccine. NIAID AIDS Vaccine Evaluation Group. AIDS. 2000 Jul 7;14(10):1365-74. doi: 10.1097/00002030-200007070-00009. PMID 10930151
- [Background] Kaslow RA, Rivers C, Goepfert P, Tang J, El Habib R, Weinhold K, Mulligan MJ. Association of HLA class I alleles with cytotoxic T-lymphocyte (CTL) responses to gag and env in recipients of ALVAC-HIV canarypox vaccines. 7th Conference on Retroviruses and Opportunistic Infections. 2000 Jan 30-Feb 2 [Poster 818]
- [Background] Zolla-Pazner S, Burda S, Belshe R, Duliege AM, Excler JL, Klein M. Prime/boost immunization of humans induces antibodies that react with many HIV-1 clades and neutralize several X4-, R5-, and dual-tropic primary isolates. Keystone Symposium, HIV Vaccine Development: Opportunities and Challenges--AIDS Pathogenesis. 1999 Jan 7-13 [J1:420]